CLINICAL TRIAL: NCT06476223
Title: Efficacy and Safety of Artificial Saliva Containing Cumin and Ginger Extract in Hemodialysis
Brief Title: Artificial Saliva Containing Cumin and Ginger Extract in Hemodialysis Patients With Xerostomia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0763/66
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial saliva containing cumin and ginger extract (Experimental): The sample will be sprayed 2 puff/time, 3 times/day, for 14 days.
  Interventions: Drug: Artificial saliva containing cumin and ginger extract
- Placebo (Placebo Comparator): The sample will be sprayed 2 puff/time, 3 times/day, for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Artificial saliva containing cumin and ginger extract — The sample will be sprayed 2 puff/time, 3 times/day, for 14 days.
  Arms: Artificial saliva containing cumin and ginger extract
Drug: Placebo — The sample will be sprayed 2 puff/time, 3 times/day, for 14 days.
  Arms: Placebo

SUMMARY:
Hemodialysis patients with xerostomia are divided into 2 groups which are group A (start with artificial saliva containing cumin and ginger extract for 2 weeks, free periods 2 weeks, then placebo for 2 weeks) and group B (start with placebo for 2 weeks, free periods 2 weeks, then artificial saliva containing cumin and ginger extract for 2 weeks). Amount of saliva (g/min), xerostomia's questionnaire, Increase of saliva score, World Health Organization Oral Mucositis Grading Scale, acid and base of saliva, quality of life's questionnaire will measure before, after using the sample for 7 and 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Hemodialysis patients with xerostomia (saliva flow rate less than 0.2 g/min)
* Hemodialysed history more than 3 months
* Be willing to participate in the study

Exclusion Criteria:

* Patients with sialolith or Sjogren's syndrome
* Uncontrolled other diseases
* Using artificial saliva for more than 2 weeks
* Taking pilocarpine and cevimeline
* Allergic to ginger, cumin, xylitol, and glycerin
* Have mucositis
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Xerostomia symptoms using Xerostomia Inventory Score | 14 days
  Patients give the score of Xerostomia Inventory questionnaire. The Xerostomia Inventory Score is graded 11 to 55 (Low score means low frequency xerostomia and high score means high frequency of xerostomia)

SECONDARY OUTCOMES:
Salivary flow rate | 14 days
  Weigh the saliva amount from the patients in 5 mins and then calculate in g/min
Amount of saliva score | 14 days
  Patients give the score of saliva amount (0 to 10, 0 means no saliva and 10 means high amount of saliva)
Quality of life score using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck 35 | 14 days
  Patients give the score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck 35. The score is graded 35 to 130 (Low score means high quality of life and high score means low quality of life)
World Health Organization Oral Mucositis | 14 days
  World Health Organization Oral Mucositis is graded 0 to 4 (0 means no mucositis to 4 means severe mucositis).
Acid and base of saliva | 14 days
  Measure acid and base of saliva using acid and base standard paper